CLINICAL TRIAL: NCT02871479
Title: A Double-Blind, Randomized, Placebo-Controlled, Safety, Tolerability, and Efficacy Trial of a Novel Botanical Drug Product Containing East Indian Sandalwood Oil (EISO) For The Treatment of Atopic Dermatitis
Brief Title: A Trial of a Botanical Drug Containing East Indian Sandalwood Oil (EISO) For Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santalis Pharmaceuticals, Inc. (Industry)
Collaborators: ClinDatrix, Inc. (Industry); Texas Dermatology and Laser Specialists (Unknown); Clinical Trials of Texas, Inc. (Other); Derm Research, PLLC (Other); Progressive Clinical Research (Other); U.S. Dermatology Partners Bryan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAN007-02
Record Dates: First submitted 2016-08-11; First posted 2016-08-18 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAN007 5% cream (Experimental): A cream containing 5% East Indian sandalwood oil (EISO).
  Interventions: Drug: SAN007 5% cream
- Placebo cream (Placebo Comparator): The vehicle cream
  Interventions: Drug: Placebo
- SAN007 10% cream (Experimental): A cream containing 10% East Indian Sandalwood Oil (EISO).
  Interventions: Drug: SAN007 10% cream

INTERVENTIONS:
Drug: SAN007 5% cream — 5% EISO in a cream formulation applied twice a day for up to 28 days.
  Other Names: Albuterpenoids; East Indian sandalwood oil (EISO)
  Arms: SAN007 5% cream
Drug: Placebo — A placebo cream containing the same components as the vehicle for the active intervention arm
  Other Names: vehicle cream
  Arms: Placebo cream
Drug: SAN007 10% cream — 10% EISO in a cream formulation applied twice a day for up to 28 days.
  Other Names: Albuterpenoids; East Indian Sandalwood Oil (EISO)
  Arms: SAN007 10% cream

SUMMARY:
This trial will be a double-blind, randomized, placebo-controlled, safety, tolerability and efficacy trial of SAN007 (5% East Indian sandalwood oil in a cream formulation) treatment regimen when administered daily for up to 28 days to patients at least 18 years of age, with atopic dermatitis.

DETAILED DESCRIPTION:
Subjects will enter the Screening Period once the informed consent/ascent and photographic consent process has been completed. Subjects with a total body surface area (BSA) of ≥2% and ≤ 15% atopic dermatitis involvement, in the treatable areas, and who meet all of the inclusion and none of the exclusion criteria will be enrolled.

Once subject eligibility is confirmed and the screening procedures completed, the subject will start the Treatment Period of the study. All enrolled subjects will receive either 5% SAN007 cream or placebo cream (randomized in a 2:1 ratio) OR 10% SAN007 cream or placebo cream (randomized in a 2:1 ratio) with the first dose applied at Visit 1 Baseline. Subjects will be instructed on how to apply the study medication twice daily for 28 days. Subjects will return to the clinic on Study Days 7,14 and 28 for study-related assessments. Subjects will receive a telephone contact from the site, on Study Days 21 and 35.

Safety will be assessed by evaluating adverse events (AEs) with respect to severity, duration, and relationship to study drug.

In addition, cutaneous tolerability will be evaluated at each visit. Tolerability evaluation will be based on subjects reporting discomfort during or immediately following application of SAN007. This will also be recorded as an AE. The study exclusion areas are not to be included in this evaluation.

Efficacy will be assessed at each study visit through the completion of the IGA, EASI and BSA calculation.

During the active treatment period, subjects will return to the study site according to the study schedule for interim assessments and recording of concomitant medication and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included in the trial if they meet all of the following criteria:

  1. Are at least 18 years of age
  2. Have atopic dermatitis, as determined by an EASI score of ≥5 and ≤50 (Hanifin, 2001)
  3. Total treatment area(s) of atopic dermatitis involvement ≥2% and ≤15% today surface area (BSA).
  4. Have atopic dermatitis that has been clinically stable for ≥ 30-days prior to the Screening Visit.
  5. Are able to obtain written informed consent/ascent in a manner approved by the Institutional Review Board and comply with the requirements of the study.
  6. Are willing to refrain from using any lotions, moisturizer, cleansers, cosmetics or creams, other than those issued as part of the study, on the target treatment areas during the treatment period.
  7. Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events.
  8. Are willing to refrain from exposure to artificial ultraviolet radiation for the duration of the study.
  9. Are willing to cover target treatment areas to avoid exposure to natural ultraviolet radiation for the duration of the study.
  10. If female of childbearing potential, must be willing to practice an acceptable form of birth control for the duration of the study. i.e. barrier method, hormone or intrauterine device.
  11. Are willing to avoid participation in any other interventional clinical trial for the duration of this study.
  12. Are willing to refrain from treating areas that are not in the defined treatment area(s), which will be excluded from the IGA assessments and BSA calculation. These areas are as follows: head, neck, soles of feet, palms of hands, axillae, or intertriginous areas.

Exclusion Criteria:

* Subjects will be excluded from the trial if they meet any of the following criteria:

  1. Have a sibling or immediate family member already participating in this trial.
  2. Currently requires and/or, in the 30 days prior to Screening, has required topical use of a medium or high potency steroid (i.e. >1%)
  3. Atopic dermatitis that, in the opinion of the investigator, is likely to stem from an allergic reaction. (i.e. contact dermatitis)
  4. Have <2% or >15% total BSA of atopic dermatitis involvement in the target treatment area(s).
  5. Have participated in any interventional clinical trial in the previous 30 days to the screening visit.
  6. Have a known sensitivity to any of the constituents of the test product including sensitivities to sandalwood oil, fragrances or any member of the Compositae family of vascular plants (e.g., sunflowers, daisies, dahlias, etc.).
  7. Have received phototherapy within the 60 days prior to Screening.
  8. Have received any systemic medication for atopic dermatitis in the past 2 months that would interfere with the evaluation of atopic dermatitis (excluding antihistamines or leukotriene inhibitors).
  9. Have a present condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
  10. Are pregnant, breast-feeding or plan to become pregnant at any point for the duration of the trial.
  11. Are not willing to practice an approved form of birth control while on the study drug for the duration of the trial. i.e. barrier method, hormone or intrauterine device.
  12. Have been treated, with prescription medication for atopic dermatitis, within 60 days prior to the Baseline visit.
  13. Have any evidence of systemic cancer, squamous cell carcinoma, basal cell carcinoma, in the last 5 years,or any other confounding skin condition.
  14. Have undergone treatments with topical atopic dermatitis drug products, other than retinoids or corticosteroids, within 14 days prior to the Baseline Visit, and for therapy containing corticosteroids or retinoids within 28 days prior to Baseline Visit.
  15. Have open sores or open lesions in the treatment area(s).
  16. Have a history of alcohol or illegal drug/substance abuse, or suspected alcohol or illegal drug/substance abuse in the past 2 years.
  17. Require greater than 2.0 mg/day inhaled or intranasal corticosteroids.
  18. Have an active infection of any kind at Visit 1 (Baseline)
  19. Have an occupation that requires ≥50% of time be spent outdoors, where prolonged exposure to ultraviolet radiation is unavoidable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Browning, MD, Principal Investigator — Texas Dermatology and Laser Specialists
Locations (5):
- United States (5):
  - DermResearch, Austin, Texas
  - J&S Sudies Pharmaceutical, Bryan, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SAN007 5% Cream | Placebo Cream | SAN007 10% Cream
Started | 36 | 24 | 11
Completed | 33 | 21 | 11
Not Completed | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAN007 5% Cream | Placebo Cream | SAN007 10% Cream | Total
Number analyzed (Participants) | 36 | 24 | 11 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (15.59) | 37.0 (13.36) | 29.6 (10.4) | 35.3 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 8 | 50
  Male | 14 | 4 | 3 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 7 | 2 | 24
  Not Hispanic or Latino | 21 | 17 | 9 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 12 | 2 | 20
  White | 27 | 11 | 8 | 46
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 | 24 | 11 | 71
Baseline EASI score [Mean (Standard Deviation); unit: units on a scale] — EASI score is used to measure the severity and extent of eczema. The index is applied to four body regions.The intensity of eczema and the percentage of the affected area are calculated for each region. The intensity of eczema is rated on a 4-point scale of 0-3.
  The four intensity scores are added up for each of the four regions to give subtotal. Each subtotal is multiplied by the body surface area represented by that region The % area affected is evaluated in 4 regions of the body.
  Each of the body area scores are multiplied by the area affected:
  EASI= C1 + C2 + C3 + C4.
  units on a scale | 6.45 (3.51) | 6.28 (4.128) | 7.41 (5.73) | 6.54 (4.074)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: Safety will be assessed by evaluating adverse events (AEs) with respect to severity, duration, and relationship to study drug.
Time Frame: 28 days
Population: The FAS group was used for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | SAN007 5% Cream | Placebo Cream | SAN007 10% Cream
Number analyzed (Participants) | 35 | 23 | 11
Participants | 7 | 5 | 1

2. Secondary Outcome: Percentage of Subjects Who Have a ≥ 50% Reduction in the Eczema Area and Severity Index (EASI) Score
Description: Percentage of subjects who have a ≥ 50% reduction in the Eczema Area and Severity Index (EASI) score at any point during the trial. Minimum value is a 0 and a maximum value is 72. Higher score denoting worse than a lower score.
Time Frame: 28 days
Population: The FAS group was used for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | SAN007 5% Cream | Placebo Cream | SAN007 10% Cream
Number analyzed (Participants) | 35 | 23 | 11
Participants | 17 | 12 | 6

ADVERSE EVENTS:
Time Frame: AE's were observed over the course of the treatment period, which was 28 days.
Arm/Group | SAN007 5% Cream | Placebo Cream | SAN007 10% Cream
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/24 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/24 | 0/11
Other Adverse Events (participants affected / at risk) | 0/36 | 2/24 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAN007 5% Cream (N=36) | Placebo Cream (N=24) | SAN007 10% Cream (N=11)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT02871479/SAP_000.pdf
  • Study Protocol (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT02871479/Prot_001.pdf